CLINICAL TRIAL: NCT00890448
Title: A Modified Case Control Study to Identify Pharmacogenomic Factors Associated With Hepatocellular Injury Following Exposure to Lapaquistat Acetate
Brief Title: Case Control Study of Pharmacogenomic Factors Associated With Hepatocellular Injury Following Exposure to Lapaquistat Acetate
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-475_310; 2008-006906-41 (Registry Identifier: EudraCT); U1111-1112-3768 (Registry Identifier: WHO); DOH-27-0410-2857 (Registry Identifier: SANCTR)
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Toxicity
Keywords: Alanine Transaminase elevation; Genetic Markers; DNA Markers
MeSH Terms: interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Pharmacogenomic whole blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lapaquistat acetate participants
  Interventions: Other: Pharmacogenomic whole blood sampling

INTERVENTIONS:
Other: Pharmacogenomic whole blood sampling — 10 mL, whole blood, one sample on Visit 2
  Other Names: TAK-475

SUMMARY:
The purpose of this study is to examine the genetic contribution to the mechanism of lapaquistat acetate- induced hepatic abnormalities.

DETAILED DESCRIPTION:
This is a modified case control study to investigate the association of genotype with phenotype in subjects who experienced alanine aminotransferase and bilirubin derangements following exposure to lapaquistat acetate.

The DNA profile of subjects who experienced significant biochemical hepatic derangement following exposure to lapaquistat acetate (cases) will be compared with a population of pre-genotyped untreated individuals (controls) from a public database. The DNA from subjects who had hepatic derangement during lapaquistat acetate studies, in the absence of exposure to lapaquistat acetate, will be stored. If data from the subjects exposed to lapaquistat acetate indicates that there is a genetic marker of interest, the stored DNA from non-exposed subjects will be assayed to further investigate the signal. One 10 mL sample of whole blood will be collected in plastic K2EDTA tube, after informed consent has been obtained.

Each subject will sign the informed consent document prior to undergoing the study-related procedure. One 10 mL sample of whole blood will be collected from each subject. Extracted DNA will be analyzed using a whole genome scan approach as well as a candidate gene approach.

ELIGIBILITY:
Inclusion Criteria:

* Has experienced an alanine aminotransferase level greater than or equal to 5 times the upper limit of normal, or concurrent elevation of alanine aminotransferase greater than or equal to 3 times the upper limit of normal and bilirubin greater than or equal to 2 times the upper limit of normal while participating in lapaquistat acetate clinical studies.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who participated in lapaquistat acetate phase 2 and phase 3 clinical studies
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Whole genome scanning using the Illumina 1M chip. | Visit 2
Whole genome scanning using the Affymetrix 500K array chip. | Visit 2
Candidate gene scanning using the Affymetrix Drug Metabolizing Enzymes and Transporter (DMET) array. | Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (19):
- United States (4):
  - Jacksonville, Florida
  - Jupiter, Florida
  - Idaho Falls, Idaho
  - Richmond, Virginia
- Córdoba, Argentina
- Canada (2):
  - Québec
  - Sainte-Foy
- Santiago, Chile
- Havírov-Šumbark, Czechia
- Oulu, Finland
- Nuremberg, Germany
- Riga, Latvia
- Groningen, Netherlands
- Gdansk, Poland
- Russia (2):
  - Moscow
  - Saratov
- Žilina, Slovakia
- Johannesburg, South Africa
- Glasgow, Scotland, United Kingdom